CLINICAL TRIAL: NCT04270318
Title: Clinical, Radiographic, and Histologic Outcome of Sodium Hypoclorite as an Antibacterial Agent Prior to Calcium Hydroxide and Mineral Trioxide Aggregate Pulpotomies in Primary Teeth
Brief Title: Sodium Hypoclorite as an Antibacterial Agent Prior to Pulpotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Merve AKCAY, Assoc. Prof., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-TEZ-07
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pulpotomy; Primary Teeth
Keywords: calcium hydroxide; mineral trioxide aggregate; sodium hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CH pulpotomy-control (Active Comparator): After hemorrhage control, pulp chamber was cleansed with physiologic saline prior the CH pulpotomy.Then, canal orifices were sealed with CH (Kalsin, Aktu, Izmir, Turkey) paste (CH powder mixed with physiologic saline). After the canal orifice dressing, the chamber was based with reinforced ZOE (IRM; Dentsply Caulk, Milford, DE) and the tooth immediately restored with a stainless steel crown (SSC; 3M ESPE, Seefeld, Germany).
  Interventions: Other: CH Pulpotomy, physiologic saline
- CH pulpotomy-NaOCl (Experimental): After hemorrhage control,pulp chamber was cleansed with 5% NaOCl for 30 s prior the CH pulpotomy. Then, canal orifices were sealed with CH (Kalsin, Aktu, Izmir, Turkey) paste (CH powder mixed with physiologic saline). After the canal orifice dressing, the chamber was based with reinforced ZOE (IRM; Dentsply Caulk, Milford, DE) and the tooth immediately restored with a stainless steel crown (SSC; 3M ESPE, Seefeld, Germany).
  Interventions: Other: CH pulpotomy, NaOCl
- MTA pulpotomy-control (Active Comparator): After hemorrhage control, pulp chamber was cleansed with physiologic saline prior the MTA pulpotomy. Then, canal orifices were sealed with MTA (ProRoot MTA; Dentsply, Tulsa, OK, USA) and a moistened cotton pellet was placed over the MTA paste to allow setting of the material. Reinforced ZOE was placed as a temporary restoration; the ZOE and the cotton pellets were removed after 24 h, and the teeth finally restored with SSCs.
  Interventions: Other: MTA Pulpotomy, physiologic saline
- MTA pulpotomy-NaOCl (Experimental): After hemorrhage control, pulp chamber was cleansed with physiologic saline prior the MTA pulpotomy. MTA NaOCl (n = 31 teeth): Pulp chamber was cleansed with 5% NaOCl for 30 s prior the MTA pulpotomy.
  Then, canal orifices were sealed with MTA (ProRoot MTA; Dentsply, Tulsa, OK, USA) and a moistened cotton pellet was placed over the MTA paste to allow setting of the material. Reinforced ZOE was placed as a temporary restoration; the ZOE and the cotton pellets were removed after 24 h, and the teeth finally restored with SSCs.
  Interventions: Other: MTA pulpotomy, NaOCl

INTERVENTIONS:
Other: CH Pulpotomy, physiologic saline — Pulp chamber was cleansed with physiologic saline for 30 s.
  Arms: CH pulpotomy-control
Other: CH pulpotomy, NaOCl — Pulp chamber was cleansed with 5 % NaOCl for 30 s.
  Arms: CH pulpotomy-NaOCl
Other: MTA Pulpotomy, physiologic saline — Pulp chamber was cleansed with physiologic saline for 30 s.
  Arms: MTA pulpotomy-control
Other: MTA pulpotomy, NaOCl — Pulp chamber was cleansed with 5 % NaOCl for 30 s.
  Arms: MTA pulpotomy-NaOCl

SUMMARY:
Aim: The aim of this study was to report the 24-Month radiographical and histological outcome on these previously reported calcium hydroxide (CH) and mineral trioxide aggregate (MTA) pulpotomies using of five percent sodium hypochlorite (NaOCl) as an antibacterial agent to clean the chamber prior to application of the pulpotomy agent.

Materials and Methods: 128 primary molars were randomly divided into two main groups according to pulpotomy material (CH/MTA) and into two sub-groups according to selected the antibacterial agent (NaOCl/physiologic saline) used in the pulpotomy procedure. After these procedures, teeth were followed radiographically for 24 months. Thirty-four successfully treated teeth whose successors roots had completed formation of at least two-thirds of their lengths were extracted for histological evaluation. Fisher's-exact test, Pearson's-chi-square test and MannWhitneyU test with Bonferroni correction were used for statistical analysis.

DETAILED DESCRIPTION:
The procedure and possible discomforts, risks, and benefits had been fully explained to the parents of the children, and informed consent forms were signed.

A total of 64 children (37 boys and 27 girls), between six to 10 years old (mean=8.2 years old) who had at least two mandibular primary molars with nearly equal carious involvement that required pulpotomy were included in the study. Following anesthesia and rubber dam isolation, the pulpotomy procedure was realized. After amputation of the coronal pulp tissue, pulpal hemorrhage was controlled using dry sterile cotton pellets under slight pressure for approximately 5 min. Four teeth were excluded from the study because of uncontrolled bleeding.

A total of 124 teeth were randomly distributed (by a coin toss) among groups representing different pulpotomy materials (CH or MTA) and cleansing agents (NaOCl or physiologic saline).

CH pulpotomy (n = 62 teeth): After hemorrhage control, two teeth in each child were randomly assigned by the toss of a coin to receive two cleansing agents, the experimental disinfecting agent 5% NaOCl (Wizard, Rehber Chemistry, Istanbul, Turkey) or the physiologic saline. CH control (n = 31 teeth): Pulp chamber was cleansed with physiologic saline prior the CH pulpotomy. CH NaOCl (n = 31 teeth): Pulp chamber was cleansed with 5% NaOCl for 30 s prior the CH pulpotomy. Then, canal orifices were sealed with CH (Kalsin, Aktu, Izmir, Turkey) paste (CH powder mixed with physiologic saline). After the canal orifice dressing, the chamber was based with reinforced ZOE (IRM; Dentsply Caulk, Milford, DE) and the tooth immediately restored with a stainless steel crown (SSC; 3M ESPE, Seefeld, Germany).

MTA pulpotomy (n = 62 teeth): As stated above, following the hemorrhage control, two cleansing agents were randomly applied to the cavity. MTA control (n= 31 teeth): Pulp chamber was cleansed with physiologic saline prior the MTA pulpotomy. MTA NaOCl (n = 31 teeth): Pulp chamber was cleansed with 5% NaOCl for 30 s prior the MTA pulpotomy. Then, canal orifices were sealed with MTA (ProRoot MTA; Dentsply, Tulsa, OK, USA) and a moistened cotton pellet was placed over the MTA paste to allow setting of the material. Reinforced ZOE was placed as a temporary restoration; the ZOE and the cotton pellets were removed after 24 h, and the teeth finally restored with SSCs.

The treatments received follow-up evaluations every six months, for 24 months, following the completion of the treatments. One examiner, who was blinded to treatment type, evaluated the teeth clinically and radiographically. At follow-up appointments, clinical success was confirmed by the absence of spontaneous pain, pathologic mobility, tenderness to percussion, swelling, fistula, or gingival inflammation. Radiographic success was considered when internal/external root resorption and periapical/furcal radiolucency was not observed. Calcific metamorphosis of the pulp was not considered a failure. The data were analyzed using Fisher's exact, McNemar, and Pearson's chi-square tests with Bonferroni correction.

Histological assessment Clinically and radiologically successful teeth -whose successors roots had completed formation of at least two thirds of their lengths- were extracted for histopathological evaluation. Following extraction, the teeth were immediately immersed in 10 % buffered formalin, embedded in paraffin, and serially sectioned through the root canals in a mesiodistal direction using a microtome to obtain sections of 5 μm in thickness. Sections were stained using hematoxylin eosin and examined under a light microscope.

ELIGIBILITY:
Inclusion Criteria:

* Each child had at least two previously untreated lower 2nd primary mandibular molars with nearly equal carious involvement that required pulpotomies but showed positive response to vitality tests (electrical pulp test and cold stimulation)
* The children were healthy and cooperative
* Moderate response to chemical and thermal stimuli.
* Teeth would be restorable with stainless steel crowns.

Exclusion Criteria:

* Signs of irreversible pulpitis (such as spontaneous pain, prolonged pain response),
* Presence of percussion or palpation,
* Pathological mobility,
* Infectious symptoms such as fistula or abscess,
* Discoloration in the clinical examination,
* Presence of radiolucency in the furcation or periodical regions thickening of the periodontal spaces
* Internal or external root resorption.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Clinical success rate of pulpotomy | Change of clinical success from baseline at 12 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of spontaneous pain, pathologic mobility, tenderness to percussion, swelling, fistula, or gingival inflammation. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Clinical success rate of pulpotomy | Change of clinical success from Baseline at 24 month
  Treatment is considered a clinical failure if one or more of the following signs are observed: Presence of spontaneous pain, pathologic mobility, tenderness to percussion, swelling, fistula, or gingival inflammation. The treatment is regarded successful if clinical evaluation does not indicate any signs of failure.
Radiographic success rate of pulpotomy | Change of radiographicsuccess from baseline at 12 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.
  success was considered when internal/external root resorption and periapical/furcal radiolucency was not observed.
Radiographic success rate of pulpotomy | Change of radiographicsuccess from baseline at 24 month
  For radiographic evaluation, the treatment is rated as a failure when one or more of the following signs are present: lesions in the furcation or periapical regions, internal or external root resorption, and thickening of the periodontal spaces. The treatment is regarded successful if radiographic evaluation does not indicate any signs of failure.
  success was considered when internal/external root resorption and periapical/furcal radiolucency was not observed.

SECONDARY OUTCOMES:
Histological success rate of indirect pulp treatment | up to 30 months (the teeth were extracted in regular exfoliation period (in which the underlying permanent tooth germ had completed 2/3 of root formation).]
  For histologic evaluation, the treatment is rated as a failure when one or more of the following signs are present: absent of the integrity of the odontoblastic layer, absent of tertiary dentin formation, presence of pulpitis, presence of fibrosis and dystrophic calcification. The treatment is regarded successful if histologic evaluation does not indicate any signs of failure.